CLINICAL TRIAL: NCT00401024
Title: Determination of the In-Tumor-Concentration of Imatinib Mesylate in Malignant Glioma After Oral Administration
Brief Title: Tumor Tissue Analysis in Patients Receiving Imatinib Mesylate for Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0623; P30CA006973 (NIH); CDR0000510133; NA_00001201 (Other: JHM IRB)
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic oligodendroglioma; adult oligodendroglioma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma; recurrent adult brain tumor; adult brain stem glioma; adult mixed glioma; adult glioblastoma; adult pilocytic astrocytoma; adult diffuse astrocytoma; adult anaplastic ependymoma; adult ependymoma; adult myxopapillary ependymoma; adult subependymoma; adult pineal gland astrocytoma; adult subependymal giant cell astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Astrocytoma; Glioblastoma; Gliosarcoma; Brain Neoplasms; Glioma; Ependymoma; Glioma, Subependymal | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Imatinib mesylate 600mg orally once a day for seven consecutive days prior to surgery with last dose taken one day prior to surgery
  Interventions: Drug: imatinib mesylate; Other: pharmacological study; Procedure: conventional surgery

INTERVENTIONS:
Drug: imatinib mesylate
Other: pharmacological study
Procedure: conventional surgery

SUMMARY:
RATIONALE: Collecting samples of tumor tissue and blood from patients with cancer to study in the laboratory may help doctors learn how patients respond to treatment.

PURPOSE: This clinical trial is looking at tumor tissue samples from patients receiving imatinib mesylate for malignant glioma to see how much imatinib mesylate is found in the tumor tissue.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy, of imatinib mesylate, in terms of achieving a therapeutic tumor:plasma concentration ratio, in patients with primary malignant glioma.

Secondary

* Correlate tumor grade (low vs high) and/or tumor enhancement on MRI with tumor concentration of this drug in these patients.,

OUTLINE: Patients receive oral imatinib mesylate once daily for 7-12 days. Patients then undergo surgical resection.

Blood and tissue samples are collected at the time of surgery and analyzed for imatinib mesylate concentration.

After completion of study treatment, patients are followed for 7 days.

PROJECTED ACCRUAL: A total of 33 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma of 1 of the following subtypes:

  * Low-grade glioma
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Glioblastoma multiforme
* Unifocal disease that is progressive or recurrent after prior radiotherapy and/or chemotherapy
* Scheduled to undergo surgical resection

  * Able to undergo maximal surgical resection of tumor mass

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Mini Mental Status Exam ≥ 15
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≥ 1.7 mg/dL
* BUN ≤ 2 times upper limit of normal (ULN)
* Transaminases ≤ 4 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for ≥ 1 month after completion of study treatment
* No other medical illness that would preclude study treatment, including any of the following:

  * Serious infection
  * Uncontrolled hypertension
  * Unstable angina pectoris
  * Uncontrolled cardiac dysrhythmia

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* At least 4 weeks since prior investigational drugs
* No more than 1 prior chemotherapy regimen
* No concurrent chemotherapy, biologic therapy, or radiotherapy
* No concurrent medications that may interact with imatinib mesylate or interfere with hepatic cytochrome P450 system

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-10-12 (Actual); Primary Completion 2008-02-04 (Actual); Study Completion 2008-11-11 (Actual)

PRIMARY OUTCOMES:
Tumor:plasma concentration ratio of imatinib mesylate | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A. Grossman, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Holdhoff M, Supko JG, Gallia GL, Hann CL, Bonekamp D, Ye X, Cao B, Olivi A, Grossman SA. Intratumoral concentrations of imatinib after oral administration in patients with glioblastoma multiforme. J Neurooncol. 2010 Apr;97(2):241-5. doi: 10.1007/s11060-009-0008-0. Epub 2009 Sep 19. PMID 19768386